CLINICAL TRIAL: NCT02174276
Title: A Phase 2, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of GS-4774 in Combination With Tenofovir Disoproxil Fumarate (TDF) for the Treatment of Subjects With Chronic Hepatitis B and Who Are Currently Not on Treatment
Brief Title: Safety and Efficacy of GS-4774 in Combination With Tenofovir Disoproxil Fumarate (TDF) for the Treatment of Participants With Chronic Hepatitis B (CHB) and Who Are Currently Not on Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-330-1401; 2014-001011-39 (EudraCT Number)
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TDF 48 weeks (Active Comparator): Participants will receive TDF for 48 weeks. After Week 48, participants will have the option to continue receiving TDF for up to 144 weeks.
  Interventions: Drug: Tenofovir disoproxil fumarate
- TDF plus GS-4774 2 YU (Experimental): Participants will receive TDF plus GS-4774 2 yeast units (YU) for 20 weeks. After Week 20, GS-4774 will be discontinued and participants will continue on TDF for an additional 28 weeks. After Week 48, participants will have the option to continue receiving TDF for up to 144 weeks.
  Interventions: Drug: Tenofovir disoproxil fumarate; Biological: GS-4774
- TDF plus GS-4774 10 YU (Experimental): Participants will receive TDF plus GS-4774 10 YU for 20 weeks. After Week 20, GS-4774 will be discontinued and participants will continue on TDF for an additional 28 weeks. After Week 48, participants will have the option to continue receiving TDF for up to 144 weeks.
  Interventions: Drug: Tenofovir disoproxil fumarate; Biological: GS-4774
- TDF plus GS-4774 40 YU (Experimental): Participants will receive TDF plus GS-4774 40 YU for 20 weeks. After Week 20, GS-4774 will be discontinued and participants will continue on TDF for an additional 28 weeks. After Week 48, participants will have the option to continue receiving TDF for up to 144 weeks.
  Interventions: Drug: Tenofovir disoproxil fumarate; Biological: GS-4774

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — TDF 300 mg tablet administered orally once daily
  Other Names: TDF; Viread®
Biological: GS-4774 — GS-4774 subcutaneous injection administered every 4 weeks for a total of 6 doses
  Arms: TDF plus GS-4774 10 YU; TDF plus GS-4774 2 YU; TDF plus GS-4774 40 YU

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, and efficacy of GS-4774 in adults with CHB and who are currently not on treatment. Participants will be randomized to receive TDF alone or GS-4774 plus TDF for 20 weeks. After Week 20, GS-4774 will be discontinued. All participants will continue on TDF and will be followed for an additional 28 weeks. Following completion of the 48 week study period, all participants will be eligible for a treatment extension for 96 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study
* Documented evidence of chronic hepatitis B virus (HBV) infection, for example, hepatitis B surface antigen (HBsAg) positive for more than 6 months
* Screening HBV DNA ≥ 2000 IU/mL
* A negative serum pregnancy test is required for females (unless surgically sterile or > 2 years post-menopausal)

Key Exclusion Criteria:

* Cirrhosis
* Inadequate liver function
* Co-infection with hepatitis C virus (HCV), HIV or hepatitis D virus (HDV)
* Received antiviral treatment for HBV within 3 months of screening
* Evidence of hepatocellular carcinoma (eg, as evidenced by recent imaging)
* Significant cardiovascular, pulmonary, or neurological disease
* Women who are pregnant or may wish to become pregnant during the course of the study
* Received solid organ or bone marrow transplant
* Received prolonged therapy with immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, interferon) within 3 months of screening
* Use of investigational agents within 3 months of screening
* Current alcohol or substance abuse judged by the investigator to potentially interfere with individual's compliance
* Receipt of immunoglobulin or other blood products within 3 months prior to enrollment
* History of demyelinating disease (Guillain-Barre), Bell's Palsy, Crohn's disease, Ulcerative colitis, or autoimmune disease
* Documented history of yeast allergy
* Known hypersensitivity to study drugs, metabolites or formulation excipients
* Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Individuals under evaluation for possible malignancy are not eligible

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-07-24 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (33):
- United States (12):
  - Stanford University Medical Center, Palo Alto, California
  - Kaiser Permanente, Sacramento, California
  - Research and Education, Inc., San Diego, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - The Queen's Medical Center, Honolulu, Hawaii
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Xiaoli Ma, PC, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
  - Kaiser Permanente, Springfield, Virginia
- Canada (6):
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Liver and Intestinal Research Center, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Toronto General Hospital-The University Health Network, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Toronto Western Hospital-The University Health Network, Toronto, Ontario
- Italy (4):
  - Aou-S.Orsola-Malpighi - Universita Degli Studi Di, Bologna
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Auckland Clinical Studies, Auckland, New Zealand
- Romania (2):
  - Dr. Victor Babes Hospital for Infectious Diseases, Bucharest
  - Institutul National de Boli Infectioase Prof.Dr. Matei Bals, Bucharest
- South Korea (8):
  - Kyungpook National University Hospital, Daegu
  - The Catholic University of Korea, Seocho
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Seoul National University College of Medicine, Seoul
  - Yonsei Universiity, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
  - The Catholic University of Korea, Yangsan

REFERENCES:
- [Result] Janssen HL, Yoon SK, Yoshida EM, Trinh HN, Rodell TC, Nguyen AH, et al. Safety and Efficacy of GS-4774 in combination with TDF in Patients with Chronic Hepatitis B not on Antiviral Medication [Abstract 231]. Hepatology AASLD Abstracts 2016;64 (Suppl S1):122A.
- [Result] Boni C, Janssen HLA, Rossi M, Yoon SK, Vecchi A, Barili V, Yoshida EM, Trinh H, Rodell TC, Laccabue D, Alfieri A, Brillo F, Fisicaro P, Acerbi G, Pedrazzi G, Andreone P, Cursaro C, Margotti M, Santoro R, Piazzolla V, Brunetto MR, Coco B, Cavallone D, Zhao Y, Joshi A, Woo J, Lau AH, Gaggar A, Subramanian GM, Massetto B, Fung S, Ahn SH, Ma X, Mangia A, Ferrari C. Combined GS-4774 and Tenofovir Therapy Can Improve HBV-Specific T-Cell Responses in Patients With Chronic Hepatitis. Gastroenterology. 2019 Jul;157(1):227-241.e7. doi: 10.1053/j.gastro.2019.03.044. Epub 2019 Mar 28. PMID 30930022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, New Zealand, and South Korea. The first participant was screened on 24 July 2014. The last study visit occurred on 30 May 2018.
Pre-assignment Details: 254 participants were screened.
Groups:
- TDF 48 Weeks: Participants received tenofovir disoproxil fumarate (TDF) 300 mg tablet orally once daily for 48 weeks during the main study. Participants had the option to continue receiving TDF 300 mg tablet orally once daily for up to 144 weeks (in optional treatment extension phase [OTEP]).
- TDF + GS-4774 2 YU: Participants received TDF 300 mg tablet orally once daily for 48 weeks + GS-4774 2 yeast units (YU) administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Participants had the option to continue receiving TDF 300 mg tablet orally once daily for up to 144 weeks (in OTEP).
- TDF + GS-4774 10 YU: Participants received TDF 300 mg tablet orally once daily for 48 weeks + GS-4774 10 YU administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Participants had the option to continue receiving TDF 300 mg tablet orally once daily for up to 144 weeks (in OTEP).
- TDF + GS-4774 40 YU: Participants received TDF 300 mg tablet orally once daily for 48 weeks + GS-4774 40 YU administered via subcutaneous injection every 4 weeks for 20 weeks (total of 6 doses). Participants had the option to continue receiving TDF 300 mg tablet orally once daily for up to 144 weeks (in OTEP).
Period: Study Treatment Phase (Weeks 1 to 48)
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Started | 27 | 57 | 56 | 55
Completed | 26 | 56 | 53 | 55
Not Completed | 1 | 1 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Period: OTEP (Weeks 48 to 144)
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Started | 26 | 54 (2 Participants completed the study treatment phase but did not continue in OTEP.) | 51 (2 Participants completed the study treatment phase but did not continue in OTEP.) | 52 (3 Participants completed the study treatment phase but did not continue in OTEP.)
Completed | 25 | 54 | 48 | 50
Not Completed | 1 | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Withdrew Consent | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- TDF 48 Weeks: Participants received TDF 300 mg tablet orally once daily for 48 weeks during the main study. Participants had the option to continue receiving TDF 300 mg tablet orally once daily for up to 144 weeks (in OTEP).
- Total: Total of all reporting groups
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU | Total
Number analyzed (Participants) | 27 | 57 | 56 | 55 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (10.3) | 46 (11.2) | 44 (9.1) | 43 (11.6) | 44 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 23 | 23 | 22 | 77
  Male | 18 | 34 | 33 | 33 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 24 | 42 | 44 | 45 | 155
  Race: White | 1 | 13 | 8 | 6 | 28
  Race: Black or African American | 2 | 2 | 2 | 3 | 9
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 27 | 54 | 56 | 55 | 192
  Ethnicity: Not Permitted | 0 | 3 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 0 | 0 | 1 | 0 | 1
  Canada | 6 | 14 | 9 | 17 | 46
  South Korea | 9 | 16 | 19 | 12 | 56
  Romania | 0 | 2 | 2 | 3 | 7
  United States | 11 | 20 | 20 | 21 | 72
  Italy | 1 | 5 | 5 | 2 | 13
Baseline Hepatitis B Surface Antigen (HBsAg) [Mean (Standard Deviation); unit: log10 IU/mL] | 3.8 (0.78) | 3.7 (0.82) | 3.7 (0.94) | 3.7 (0.80) | 3.7 (0.84)
Baseline Hepatitis B Virus (HBV) DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.0 (1.64) | 5.8 (1.99) | 5.8 (1.97) | 6.0 (1.80) | 5.9 (1.88)
Hepatitis B Envelope Antigen (HBeAg) Status at Baseline [Count of Participants; unit: Participants]
  Positive | 10 | 22 | 23 | 21 | 76
  Negative | 17 | 35 | 33 | 34 | 119
Baseline Alanine Aminotransferase (ALT) Category [Count of Participants; unit: Participants] — Upper limit of normal (ULN) for ALT was defined as 19 U/L for women and 30 U/L for men.
  Participants
    ≤ ULN | 6 | 15 | 21 | 12 | 54
    > ULN | 21 | 42 | 35 | 43 | 141

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Serum HBsAg From Baseline to Week 24
Description: The change from baseline to Week 24 in HBsAg was analyzed using a mixed effect model for repeated measures (MMRM). The model included treatment groups, ALT levels (> ULN or ≤ ULN) at baseline, HBeAg status (positive or negative) at baseline, HBsAg level at baseline, visit and treatment-by-visit interaction as fixed effects and visit as a repeated measurement. Estimated least square means of treatment effects are presented with the 95% confidence intervals (CIs).
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set (all participants who were randomized and received at least 1 dose of study drug) with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 26 | 57 | 54 | 55
log10 IU/mL | -0.079 [-0.192 to 0.035] | -0.096 [-0.174 to -0.018] | -0.016 [-0.095 to 0.064] | -0.135 [-0.215 to -0.055]
Statistical Analysis 1: Comparison: TDF 48 Weeks vs TDF + GS-4774 2 YU; The null hypotheses was that the mean change from baseline in serum HBsAg in each of the TDF + GS-4774 groups was equal to the mean change from baseline in serum HBsAg in the TDF only group. Each null hypothesis was tested against the 2-sided alternative hypothesis that the mean change from baseline in serum HBsAg was not equal between each of the respective GS-4774 dose groups and the TDF only group; Test type: Superiority — Estimated differences in treatment effects between GS-4774 treatment groups and the TDF only group at Week 24 are presented with the 95% CIs and unadjusted P-values; p = 0.805, Mixed-Effect Model for Repeated Measures; Least Square Mean Difference = -0.017, 95% CI 2-sided [-0.155 to 0.120]
Statistical Analysis 2: Comparison: TDF 48 Weeks vs TDF + GS-4774 10 YU; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.370, Mixed-Effect Model for Repeated Measures; Least Square Mean Difference = 0.063, 95% CI 2-sided [-0.075 to 0.202]
Statistical Analysis 3: Comparison: TDF 48 Weeks vs TDF + GS-4774 40 YU; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.426, Mixed-Effect Model for Repeated Measures; Least Square Mean Difference = -0.056, 95% CI 2-sided [-0.194 to 0.082]

2. Secondary Outcome: Mean Change in HBsAg From Baseline to Week 12
Description: The change from baseline to Week 12 in HBsAg was analyzed using a MMRM. The model included treatment groups, ALT levels (> ULN or ≤ ULN) at baseline, HBeAg status (positive or negative) at baseline, HBsAg level at baseline, visit and treatment-by-visit interaction as fixed effects and visit as a repeated measurement. Estimated least square means of treatment effects are presented with the 95% CIs.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 55 | 54 | 54
log10 IU/mL | -0.060 [-0.165 to 0.044] | -0.061 [-0.133 to 0.011] | -0.012 [-0.086 to 0.061] | -0.095 [-0.168 to -0.021]

3. Secondary Outcome: Mean Change in HBsAg From Baseline to Week 48
Description: The change from baseline to Week 48 in HBsAg was analyzed using a MMRM. The model included treatment groups, ALT levels (> ULN or ≤ ULN) at baseline, HBeAg status (positive or negative) at baseline, HBsAg level at baseline, visit and treatment-by-visit interaction as fixed effects and visit as a repeated measurement. Estimated least square means of treatment effects are presented with the 95% CIs.
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 56 | 53 | 55
log10 IU/mL | -0.145 [-0.272 to -0.017] | -0.136 [-0.225 to -0.048] | -0.086 [-0.176 to 0.004] | -0.165 [-0.254 to -0.075]

4. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 24
Description: HBsAg loss was defined as qualitative HBsAg test changing from positive at baseline to negative at any postbaseline visit within the targeted time window.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Percentage of Participants With HBsAg Loss at Week 48
Description: as for outcome 4
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 24
Description: HBsAg loss was defined as qualitative HBsAg test changing from positive at baseline to negative at any postbaseline visit within the targeted time window. HBsAg loss and seroconversion was defined as qualitative HBsAb result changing from negative at baseline to positive at any postbaseline visit and the participant must have achieved HBsAg loss within the targeted time window.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With HBsAg Loss and HBsAg Seroconversion at Week 48
Description: as for outcome 6
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With a ≥ 0.5 Log10 IU/mL or a ≥ 1.0 Log10 IU/mL Decline in HBsAg at Week 12
Description: HBsAg with a ≥ 0.5 or ≥ 1.0 log10 IU/mL decline was defined as ≥ 0.5 or ≥ 1.0 decline from baseline in log10 IU/mL serum HBsAg at any postbaseline visit within the targeted time window.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants
  ≥ 0.5 and < 1.0 log10 IU/mL Decline | 3.7 | 3.5 | 1.8 | 5.5
  ≥ 1.0 and < 2.0 log10 IU/mL Decline | 0.0 | 3.5 | 0.0 | 0.0
  ≥ 2.0 log10 IU/mL Decline | 0.0 | 0.0 | 0.0 | 1.8

9. Secondary Outcome: Percentage of Participants With a ≥ 0.5 Log10 IU/mL or a ≥ 1.0 Log10 IU/mL Decline in HBsAg at Week 24
Description: as for outcome 8
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants
  ≥ 0.5 and < 1.0 log10 IU/mL Decline | 0.0 | 1.8 | 1.8 | 7.3
  ≥ 1.0 and < 2.0 log10 IU/mL Decline | 0.0 | 5.3 | 0.0 | 1.8
  ≥ 2.0 log10 IU/mL Decline | 0.0 | 0.0 | 0.0 | 1.8

10. Secondary Outcome: Percentage of Participants With a ≥ 0.5 Log10 IU/mL or a ≥ 1.0 Log10 IU/mL Decline in HBsAg at Week 48
Description: as for outcome 8
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants
  ≥ 0.5 and < 1.0 log10 IU/mL Decline | 11.1 | 1.8 | 7.1 | 7.3
  ≥ 1.0 and < 2.0 log10 IU/mL Decline | 0.0 | 5.3 | 1.8 | 1.8
  ≥ 2.0 log10 IU/mL Decline | 0.0 | 0.0 | 0.0 | 1.8

11. Secondary Outcome: Percentage of Participants With HBeAg Loss at Week 24
Description: HBeAg loss was defined as qualitative HBeAg test changing from positive at baseline to negative at any postbaseline visit within the targeted time window.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with HBeAg positive at baseline were analyzed. The missing equals failure approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 10 | 22 | 23 | 21
percentage of participants | 0.0 | 0.0 | 4.3 | 0.0

12. Secondary Outcome: Percentage of Participants With HBeAg Loss at Week 48
Description: as for outcome 11
Time Frame: Baseline to Week 48
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 10 | 22 | 23 | 21
percentage of participants | 0.0 | 4.5 | 8.7 | 9.5

13. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With HBeAg Loss and HBeAg Seroconversion at Week 24
Description: HBeAg loss was defined as qualitative HBeAg test changing from positive at baseline to negative at any postbaseline visit within the targeted time window. HBeAg loss and seroconversion was defined as qualitative HBeAb result changing from negative at baseline to positive at any postbaseline visit and the participant must have achieved HBeAg loss within the targeted time window.
Time Frame: Baseline to Week 24
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 10 | 22 | 23 | 21
percentage of participants | 0.0 | 0.0 | 4.3 | 0.0

14. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With HBeAg Loss and HBeAg Seroconversion at Week 48
Description: as for outcome 13
Time Frame: Baseline to Week 48
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 10 | 22 | 23 | 21
percentage of participants | 0.0 | 0.0 | 4.3 | 9.5

15. Secondary Outcome: Percentage of Participants With HBV DNA < Lower Limit of Quantification (LLOQ) at Week 24
Description: The LLOQ was defined as 20 IU/mL.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. The missing equals excluded approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 26 | 56 | 53 | 55
percentage of participants | 50.0 | 58.9 | 58.5 | 63.6

16. Secondary Outcome: Percentage of Participants With HBV DNA < LLOQ at Week 48
Description: The LLOQ was defined as 20 IU/mL.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. The missing equals excluded approach was used.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 56 | 54 | 55
percentage of participants | 70.4 | 69.6 | 69.2 | 76.4

17. Secondary Outcome: Percentage of Participants Experiencing Virologic Breakthrough at Week 24
Description: Virologic breakthrough was defined as HBV DNA ≥ 69 IU/mL after having been < 69 IU/mL, or having had ≥ 1.0 log10 increase in HBV DNA from nadir. Two consecutive visits that met the definition were required for a participant to be classified as having had virologic breakthrough.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants | 0.0 | 1.8 | 1.8 | 0.0

18. Secondary Outcome: Percentage of Participants Experiencing Virologic Breakthrough at Week 48
Description: Virologic breakthrough was defined as HBV DNA ≥ 69 IU/mL after having been < 69 IU/mL, or a ≥ 1.0 log10 increase in HBV DNA from nadir. Two consecutive visits that met the definition were required for a participant to be classified as having had virologic breakthrough.
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 27 | 57 | 56 | 55
percentage of participants | 3.7 | 5.3 | 5.4 | 0.0

19. Secondary Outcome: Number of Participants With Drug-Resistance Mutations at Week 48 or at the Last Visit Available
Description: Resistance surveillance analysis was conducted at Week 48 or Early Discontinuation (with at least 24 weeks of exposure to TDF) for any participants who met inclusion criteria (HBV DNA ≥ 69 IU/mL). Drug-resistant mutation status was assessed using HBV polymerase/ reverse transcriptase (pol/RT) population sequencing.
Time Frame: Baseline to Week 48
Population: Participants with at least 24 weeks of exposure to TDF and with HBV DNA ≥ 69 IU/mL at Week 48 or Early Discontinuation were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
Number analyzed (Participants) | 5 | 12 | 13 | 8
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to last dose date (maximum exposure: 3 years); All-Cause Mortality: First dose date up to 3 years
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | TDF 48 Weeks | TDF + GS-4774 2 YU | TDF + GS-4774 10 YU | TDF + GS-4774 40 YU
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/57 | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/27 | 1/57 | 1/56 | 1/55
Other Adverse Events (participants affected / at risk) | 12/27 | 41/57 | 50/56 | 53/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TDF 48 Weeks (N=27) | TDF + GS-4774 2 YU (N=57) | TDF + GS-4774 10 YU (N=56) | TDF + GS-4774 40 YU (N=55)
Meningitis tuberculous (Infections and infestations) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDF 48 Weeks (N=27) | TDF + GS-4774 2 YU (N=57) | TDF + GS-4774 10 YU (N=56) | TDF + GS-4774 40 YU (N=55)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 6 | 10 | 11
Asthenia (General disorders) | 0 | 1 | 1 | 3
Chills (General disorders) | 0 | 2 | 6 | 9
Fatigue (General disorders) | 5 | 10 | 21 | 22
Influenza like illness (General disorders) | 0 | 3 | 3 | 1
Injection site erythema (General disorders) | 0 | 14 | 20 | 34
Injection site induration (General disorders) | 0 | 4 | 5 | 18
Injection site oedema (General disorders) | 0 | 0 | 2 | 4
Injection site pain (General disorders) | 0 | 16 | 32 | 45
Injection site pruritus (General disorders) | 0 | 4 | 18 | 18
Injection site reaction (General disorders) | 0 | 0 | 4 | 0
Injection site swelling (General disorders) | 0 | 9 | 11 | 22
Pain (General disorders) | 0 | 1 | 3 | 4
Pyrexia (General disorders) | 1 | 3 | 1 | 7
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 3 | 5
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 9
Sinusitis (Infections and infestations) | 0 | 2 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 13 | 22
Headache (Nervous system disorders) | 2 | 9 | 17 | 20
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 8 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 1 | 5 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years